CLINICAL TRIAL: NCT02959710
Title: A Phase 1, Pilot, Single-Dose, 3-Way Crossover Study to Compare the Pharmacokinetics of AC-1204 Mixed in Water, AC-1202 Mixed in Water, and AC-1202 Mixed in Ensure® on Ketone Body Production
Brief Title: Evaluation of PK of AC-1204 Mixed in Water, AC-1202 Mixed in Water, and AC-1202 Mixed in Ensure® on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-16-013_BE
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Healthy volunteers; AC-1202; AC-1204; Pharmacokinetic; ketone body
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): AC-1204 mixed in water, AC-1202 mixed in water, AC-1202 mixed in Ensure®
  Interventions: Drug: AC-1204 mixed in water; Drug: AC-1202 mixed in water; Drug: AC-1202 mixed in Ensure®
- Group 2 (Experimental): AC-1204 mixed in water, AC-1202 mixed in water, AC-1202 mixed in Ensure®
  Interventions: Drug: AC-1204 mixed in water; Drug: AC-1202 mixed in water; Drug: AC-1202 mixed in Ensure®
- Group 3 (Experimental): AC-1204 mixed in water, AC-1202 mixed in water, AC-1202 mixed in Ensure®
  Interventions: Drug: AC-1204 mixed in water; Drug: AC-1202 mixed in water; Drug: AC-1202 mixed in Ensure®

INTERVENTIONS:
Drug: AC-1204 mixed in water — 40 g AC-1204 (shaken in 240 mL of water) at Hour 0 on Day 1
Drug: AC-1202 mixed in water — 60 g AC-1202 (shaken in 240 mL of water) at Hour 0 on Day 1
Drug: AC-1202 mixed in Ensure® — 60 g AC-1202 (shaken in approximately 8 oz [237 mL of Ensure® Original] at Hour 0 on Day 1)

SUMMARY:
To compare serum ketone body (i.e., total ketones, β hydroxybutyrate, and estimate of acetoacetate) levels after single dose administration of AC-1204 mixed in water, AC-1202 mixed in water and AC-1202 mixed in Ensure®.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male 18 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to Day -1 of Period 1 and throughout the study.
3. Body mass index (BMI) ≥ 20.0 and ≤ 30.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. At screening, subjects must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) < the upper limit of normal and triglyceride levels must be < 250 mg/dL.
5. A non vasectomized subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to Day -1 of Period 1. A subject who has been vasectomized less than 4 months prior to Day -1 of Period 1 must follow the same restrictions as a non vasectomized male).
6. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to Day -1 of Period 1.
5. History or presence of galactosemia or hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, milk, palm or coconut oil, or soy.
6. History or presence of diverticular disease, ulcers, inflammatory bowel disease or recurrent diarrhea or gout.
7. Positive urine drug or alcohol results at screening or check in.
8. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
9. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
10. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
11. QTcF interval is >460 msec or subject has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
12. Estimated creatinine clearance ≤80 mL/min at screening.
13. Unable to refrain from or anticipates the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to Day -1 of Period 1 and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
14. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to Day -1 of Period 1 and throughout the study.
15. Is lactose intolerant.
16. Is unable to complete the meal prior to Hour 0 on Day -1 of Period 1 and prior to dosing on Day 1 of Period 1.
17. Subject consumed grapefruit or Seville oranges within 14 days prior to Day -1 of Period 1.
18. Donation of blood or significant blood loss within 56 days prior to Day -1 of Period 1.
19. Plasma donation within 7 days prior to Day -1 of Period 1.
20. Participation in another clinical study within 28 days prior to Day -1 of Period 1. The 28 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day -1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
total ketones AUC0-t | 0-24 hours
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
total ketones AUC0-inf | 0-24 hours
  The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable serum concentration to the elimination rate constant.
total ketones AUC%extap | 0-24 hours
  Percent of AUC0-inf extrapolated, represented as (1 - AUC0-t/AUC0-inf)*100
total ketones Cmax | 0-24 hours
  Maximum observed concentration
total ketones Kel | 0-24 hours
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., there or more non-zero serum concentrations)
total ketones T 1/2 | 0-24 hours
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
total ketones Tmax | 0-24 hours
  Time to reach Cmax. If the value occurs at more than one time points, Tmax is defined as the first time point with this value
β hydroxybutyrate AUC0-t | 0-24 hours
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
β hydroxybutyrate AUC0-inf | 0-24 hours
  The area under the concentration time curve from time 0 extrapolated to infinity. AUC0inf is calculated as the sum of AUC0t plus the ratio of the last measurable serum concentration to the elimination rate constant.
β hydroxybutyrate AUC%extap | 0-24 hours
  Percent of AUC0-inf extrapolated, represented as (1 AUC0t/ AUC0inf)* 100
β hydroxybutyrate Cmax | 0-24 hours
  Maximum observed concentration
β hydroxybutyrate Kel | 0-24 hours
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more nonzero serum concentrations)
β hydroxybutyrate T 1/2 | 0-24 hours
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
β hydroxybutyrate Tmax | 0-24 hours
  Time to reach Cmax. If the value occurs at more than one time point, Tmax is defined as the first time point with this value
estimate of acetoacetate AUC0-t | 0-24 hours
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
estimate of acetoacetate AUC0-inf | 0-24 hours
  The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable serum concentration to the elimination rate constant.
estimate of acetoacetate AUC%extap | 0-24 hours
  Percent of AUC0-inf extrapolated, represented as (1 - AUC0-t/AUC0-inf)* 100
estimate of acetoacetate Cmax | 0-24 hours
  Maximum observed concentration
estimate of acetoacetate Kel | 0-24 hours
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-square regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero concentrations)
estimate of acetoacetate T 1/2 | 0-24 hours
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
estimate of acetoacetate Tmax | 0-24 hours
  Time to reach Cmax. If the value occurs at more than one time point, Tmax is defined as the first time point with this value

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Hunsaker, D.O., Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States